CLINICAL TRIAL: NCT04747340
Title: Clinical Effectiveness of Training for Awareness Resilience and Action (TARA) Compared to Standard Treatment for Adolescents and Young Adults With Depression, a Pragmatic Multi-center Randomised Controlled Superiority-trial
Brief Title: Clinical Effectiveness of TARA Compared to Standard Treatment for Adolescents and Young Adults With Depression
Acronym: TARA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Västerbotten County Council, Sweden (Other Government); Västernorrland County Council, Sweden (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TARA
Record Dates: First submitted 2021-01-29; First posted 2021-02-10 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-04

CONDITIONS: Depression in Adolescence; Depressive Disorder; Dysthymia and Chronic Depression
Keywords: young people; RCT; yoga; cognitive behavioural therapy; selective serotonin reuptake inhibitor; psychotherapy; biological markers; antidepressant; meditation; Magnetic resonance imaging; Emotion regulation
MeSH Terms: conditions — Depressive Disorder; Dysthymic Disorder; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Randomization stratified by center.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training for Awareness, Resilience and Action (TARA) (Experimental): 12 weekly online sessions, each 90 minutes, 6 participants/group. For participants <18 years at CAP, parents/legal guardians will participate in parts of the sessions. Manual-based: Session 1: Introducing group members; establishing guidelines; investigating attitudes and previous experiences, introducing contemplative practices. All sessions: participants sit on yoga mats. Facilitators open and briefly check-in. Participants are guided through a breathing practice, yoga-based movement (a flow of positions synchronized with the breath) and then a meditation focusing primarily on interoceptive and sensory awareness. After a short break, a psychoeducational presentation is held followed by group exercises and discussions. The sessions conclude with feedback and questions regarding the practice, followed by a description of the home practice for the coming week. Finally, participants gather their attention and have the opportunity to express their reflections and current state.
  Interventions: Behavioral: Training for Awareness Resilience and Action (TARA)
- Standard Treatment (Active Comparator): Standard treatment (ST) as given at each participating study site. ST is based on the health practitioners' knowledge, experience, current guidelines and both the practitioners' and participants' preferences. For young people with depression The Swedish National Board of Health and Welfare recommends social support and psychoeducation (as first priority), Selective Serotonin reuptake inhibitors (as second priority) and cognitive behavioral therapy (as second priority). These recommendations are generally followed and given as stand-alone treatment or in different combinations. In our study we have no control over which of these treatments are given in the ST-arm, nor the combination or timing of them. To obtain data on what treatment has been given in the ST-arm we will go through the individual medical records of all participants at the conclusion of data collection.
  Interventions: Other: Standard treatment

INTERVENTIONS:
Behavioral: Training for Awareness Resilience and Action (TARA) — See arm-description
  Arms: Training for Awareness, Resilience and Action (TARA)
Other: Standard treatment — See arm-description
  Arms: Standard Treatment

SUMMARY:
Depressive Disorders constitute an increasing global health concern and available treatments for young people have not been sufficiently effective in haltering this trend. The novel group treatment program "Training for Awareness, Resilience, and Action" (TARA) was developed to target specific mechanisms based on neuroscientific findings in adolescent depression. TARA is framed within the National Institute of Mental Health's Research Domain Criteria and has documented feasibility and preliminary efficacy in adolescents with depression.

In this study, young people (age: 15-22) with depression will be recruited from specialized Child and Adolescent Psychiatry and Youth Clinics and randomized to receive either TARA or Standard Treatment (ST) until n=67 is reached in each arm. Outcome measures will be obtained before randomization (T0), 6 weeks after treatment start (T0.5), at 3- and 6 months follow-up (T1, T2). The primary outcome measure is Reynold's Adolescent Depression Scale (RADS-2) score at T1. Secondary outcome measures are RADS-2-score at T2, clinician depression rating with Children's Depression Rating Scale, Revised at T1,and self-rated anxiety with Multidimensional Anxiety Scale for Children, 2nd ed. at T1 and T2.

Other outcomes include heart rate variability and systemic bioindicators for depression from blood and hair. Data collected from subgroups within the study will include: brain magnetic resonance imaging and accelerometry. Qualitative interviews will be performed to reach a more comprehensive understanding of the subjective experience of being depressed and to what extent treatment adequately addresses this experience. A 2-year follow-up (T3) will be performed and presented separately.

The study will be the first Randomized Controlled Trial to examine the clinical effectiveness of TARA compared to ST for young people with depression. The investigators hypothesize that (1) TARA will result in greater reduction of depression symptoms compared to ST and that group differences will be maintained or increased at T2, (2) the treatment effect of TARA will be mediated by improved emotion regulation, sleep, and psychological flexibility, (3) bioindicators for depression will improve more in the TARA-arm compared to the ST-arm, (4) it will be possible/meaningful to explore the contextual factors perceived to drive the depression onset and maintenance, and the extent to which the different treatments address these factors.

DETAILED DESCRIPTION:
The primary aim of this study is to investigate the clinical effectiveness of TARA in treating depression in adolescents and young adults by using a Randomized Controlled Trial (RCT)-design, with an active control group based on standard treatment (ST) for depression in Child and Adolescent Psychiatry (CAP) and Youth Clinics (YC). Secondary aims are: 1. to identify potential mediating effects of improved emotion regulation, sleep and psychological flexibility on the treatment effect of TARA, 2. Investigate the effects the two treatment-arms on bioindicators for depression, 3. Increase the understanding of the subjective experience of depression onset and to what extent the treatments addressed what is perceived to drive the onset and maintenance of depression.

The study is designed as a partially nested multicenter parallel-group RCT with two treatment arms: 1) TARA and 2) ST, including but not limited to anti-depressive medication such as selective serotonin reuptake inhibitors (SSRIs) and cognitive behavioral therapy. Participants are randomized to one of the two treatment arms, both delivered via the local CAP and YC unit where the participants are being either referred to, are wait-listed or treated. The study is planned in accordance with the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT) and will be analyzed and reported in accordance with the recommendations in consolidated standards of reporting trials (CONSORT).

Participants and procedures

Recruitment, treatment and data collection will be conducted in three cities in Northern Sweden, each with 1-2 centers. Several centers will be included step-wise in the RCT, until a sufficient recruitment capacity has been reached. Before including a new center the implementation of Good Clinical Practice-guide-lines, a clinical research infrastructure and the training of study-staff must be satisfactory and a pilot trial will have been conducted at each site to show feasibility. The investigators intend to recruit participants from the Child- and adolescent psychiatry (CAP) specialized outpatient academic unit and the youth outpatient community clinic (YC) in the university city Umeå (population 89 000), CAP and YC in Skellefteå (population 36 000) and CAP in Örnsköldsvik (population 33 000). The CAP unit in Sundsvall (population 55 000) is also prepared for participation, this center will be activated only if needed to maintain recruitment pace. Depending on the general recruitment rate and the feasibility of implementation of the study protocol at the different sites, one or several of the sites may be omitted.

Adolescents and young adults (15-22 years of age) with depression will be recruited to the RCT. In this study depression is defined as having a diagnosis of major depressive disorder (MDD) or persistent depressive disorder (PDD) according to DSM 5 (dysthymia in DSM-IV) or a clinician depression rating >40 using Children's Depression Rating Scale - Revised (CDRS-R). The recruitment is done through three possible pathways: 1) at the time of an incoming referral, 2) by clinical staff who recruit potential participants at their first clinical visit, from those wait-listed for treatment, or during ongoing standard treatment and 3) by participants responding to flyers posted in the local waiting-rooms and at the student health clinic at the University of Umeå.

Those who show interest in participating in the study after having received introductory information, will be provided more detailed information over the phone. At that time initial assessment for eligibility will also be performed. Further eligibility-screening is then performed online and in person (see inclusion and exclusion criteria). The decision to include a participant in the study will be made by a study-clinician on the basis of the eligibility criteria and the final decision in case of uncertainty will be made by the PI.

Before final inclusion, participants will provide written informed consent. In addition, parents/legal guardians will provide written informed consent for participants that are <18 years old. Study participation is voluntary and can be cancelled by the participant at any time.

Participants randomized to TARA who are taking antidepressant medication with maintained depressive symptoms will be offered support from a child psychiatrist to discontinue their medication over a period of 2-4 weeks and start TARA as a stand-alone treatment. Those who prefer to continue their antidepressant medication and those who require more extensive tapering regimens will still be included in the study, enter treatment as allocated and be analyzed according to the intention to treat design.

All ST will take place at the local CAP and YC units and/or be delivered online. Any worsening of symptoms during the ST will be handled by the clinic according to their standard procedures. TARA will be delivered as an online group-intervention and routines for handling potential increase of depression symptoms during TARA are explained in detail in the study protocol.

Assessment procedure

At baseline, before inclusion, self-report of sociodemographic background, social support, dissociative symptoms and adverse childhood events is completed.

After inclusion and before randomization (T0), at 3 months (T1), at 6 months (T2) and at 2 years (T3) from T0 additional self-report questionnaires are completed, for details see outcome measures. Clinician rating of depression symptom severity and global level of functioning is conducted at T0 and T1. Blood and hair samples are collected and heart rate variability (HRV) is measured at T0 and T1.

For a subgroup of randomly selected participants from both study arms in the Umeå YC/CAP-populations a 2-3 weeks of accelerometry will also be carried out at T0, 6 weeks into the study (T0,5) and at T1. MRI data acquisition will be performed at T0 and T1 in approximately n=22 randomly selected participants from each study arm from the Umeå YC/CAP-populations. MRI data acquisition will not start at the beginning of the study but will be initiated at a later time.

The TARA-participants will provide brief self-assessment and session-evaluation at the beginning and end of each session. Additionally, to evaluate mediation effects of emotion regulation, sleep and psychological flexibility three self-report scales will be administered halfway through the TARA-treatment.

Participants who do not show up for data collection will be reminded by the research team through email and/or telephone contact.

Randomization

When 6 eligible participants have been recruited at a study-site, these participants will all undergo T0 assessments within a period of 2 weeks. Next, the participants will be randomized as a group to one of the two study arms in a 1:1 allocation ratio, by a computer-generated allocation sequence using permuted blocks and stratification for center. Block sizes will vary randomly between 2 and 4 and the first value on the randomization list at each center will be discarded at random with 50% probability to reduce the risk of breaking the allocation concealment. Randomization will continue until n=67 has been reached in each arm. Codes will be used to increase information confidentiality and participant anonymity. Treatment allocation will be performed on the basis of these codes, by a different team at the Umeå University clinical research center (CRC). The CRC will not release the randomization results until the participants have been recruited into the trial and all baseline and T0 assessments have been completed. The process will thus be separate from the patient enrolment process at the clinics. Participants, TARA-facilitators and standard treatment personnel cannot be blind to treatment allocation, but clinical outcome-assessors and statistical analysts will be blinded.

Analysis

Data from the pilot-groups at each site will be analyzed and presented separately.

For the RCT, the analyses will be performed after the last participant is out and data collection at T2 is complete. No interim analyses will be conducted. Descriptive statistics will be reported using standard measures and the baseline characteristics of the included participants will be reported per randomization group in a baseline table.

All randomized participants will be included in the main analysis that will be performed according to intention to treat. The primary outcome RADS-2 total raw-score at 3 months follow up (T1) aims to investigate the differences between the two treatment arms in reduction of depressive symptoms and will be analyzed using mixed effects modelling to account for the clustering caused by partial nesting. The main mixed effects model will include fixed effects for treatment allocation, RADS-2-score at T0, age-group (dichotomous, 15-17 and 18-22 years old), study site and sex. The clustering effect will be modelled using a random intercept for each intervention group.

Superiority will be concluded if 95% confidence intervals are not overlapping between the two study-arms. Additionally, a non-inferiority margin is defined as a RADS-2 total raw-score difference of 8 points. The investigators consider this to be the maximal clinically acceptable difference in light of the other potential benefits of TARA. If superiority is not demonstrated, additional specific equivalence- and non-inferiority analyses will be performed. Since participants who withdraw or drop out may tend to have a lack of response, using the full analysis set is likely to be biased toward demonstrating non-inferiority. Therefore, a per-protocol population (defined in the study protocol) will be used in this analysis. Additionally, to avoid making biased conclusions based on the per-protocol population the analysis will also be performed on the intention to treat population and non-inferiority will be concluded if the analyses reach similar results.

Participants who do not show up for T0 assessment will not be randomized and will be considered external dropouts. Participants who complete T0-assessment and drop out before randomization will also be considered external dropouts. Participants who are randomized but do not show up for treatment or show up but do not complete the allocated treatment will be considered internal dropouts and will be included in the analysis. All participants lost to follow-up will be contacted and asked about the reason for the drop-out. This will enable a comparison between the study arms regarding the reasons for drop-out and an examination of potential sources of bias in attrition.

Additional sensitivity analyses will be performed on the primary outcome to test the robustness of findings.

Secondary outcome variables will be analyzed by using similar mixed effects models as for the primary outcome, and adjusting for the T0-value for each respective outcome. Time-point (T0, T1, T2) and the allocation by time interaction will be included as fixed effects in these models.

Time plan

Recruitment for the RCT has started. The final data collection at T2 is estimated to be completed in 2025.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient at the CAP or YC unit
* The criteria for a diagnosis Major Depressive Disorder (MDD) or Persistent Depressive disorder (PDD)/dysthymia according to the Diagnostic and Statistical Manual of Mental Disorders (DSM) IV or 5 are fulfilled. The clinical diagnosis will be validated during the screening process using the Mini International Neuropsychiatric Interview (M.I.N.I.)/Mini-International Neuropsychiatric Interview for Children and Adolescents (M.I.N.I-kid). If a diagnosis of MDD or PDD/dysthymia is not conclusive a cut-off of 40 or above on the Children's' Depression Rating Scale - Revised will be used for inclusion.
* For patients in specialist child- and adolescent psychiatry clinics below the age of 18 one parent/ legal guardian must be available and agree to participate in parts of the sessions in case the individual is randomized to the TARA-arm.

Exclusion Criteria:

1. One or several severe psychiatric co-morbid diagnoses that may interfere with or hinder group participation, including: intellectual development disorder, severe autism spectrum disorder, psychotic disorder, bipolar disorder, severe anorexia nervosa, substance use disorders, acute posttraumatic stress disorder (PTSD) and severe dissociative syndromes.
2. One or several psychiatric symptoms or behavioral problems that may interfere with or hinder group participation including:

   * Severe self-harming behavior
   * Acute suicidality, including a reported suicide attempt in the last 6 months or hospitalization for suicidality in the last 6 months
   * Disabling dissociative symptoms or > 6 points as mean item score on the Adolescent Dissociative Experiencing Scale.
   * Frequent use of recreational drugs (a urine drug screen will be performed at baseline and if positive a second test has to be negative for inclusion)
   * Reports of manic or hypomanic symptoms during the last year
3. A first degree relative with bipolar disorder (a first episode of MDD may be an incipient bipolar disorder which is not the treatment target for TARA).
4. On-going trauma, neglect, abuse or domestic violence or destabilizing legal process.
5. Pregnancy
6. Non-fluency in oral and written Swedish since the TARA groups are held in Swedish and assessment forms are in Swedish

Note:

Other psychiatric comorbidities such as attention deficit hyperactivity disorder (ADHD), anxiety, high functioning autism spectrum disorder and mild to moderate eating disorders are not considered exclusion criteria.

Accidental findings of biochemical anomalies will not be considered exclusion criteria and medical conditions will be referred for appropriate treatment.

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 136 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Reynold's Adolescent Depression Scale 2nd edition | 3 month follow-up
  Self report. Total raw-score. Raw score range is 30-120 and higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Reynold's Adolescent Depression Scale 2nd edition | 6 month follow-up
  Self report. Total raw-score. Raw score range is 30-120 and higher scores mean a worse outcome.
Children's Depression Rating Scale - Revised | 3 month follow-up
  Clinician rating. Raw score range is 17-113 and higher scores mean a worse outcome.
Multidimensional Anxiety Scale for Children | 3 month follow-up and 6 month follow-up
  Self-report. Raw score range is 0-117 and higher scores indicate a worse outcome.

OTHER OUTCOMES:
Reynold's Adolescent Depression Scale 2nd edition | 2-year follow-up
  Self-report. Total raw-score. Raw scores range is 30-120 and higher scores mean a worse outcome.
Multidimensional Anxiety Scale for Children | 2-year follow-up
  Self-report. Raw score range is 0-117 and higher scores indicate a worse outcome.
Insomnia Severity Index | 3 month follow-up, 6 month follow-up and 2-year follow-up
  Self-report. Raw score range is 0-28 and higher scores indicate a worse outcome.
Perceived Stress Scale | 3 month follow-up, 6 month follow-up and 2-year follow-up
  Self-report. Raw score range is 0-40 and higher scores indicate a worse outcome.
Avoidance and Fusion Questionnaire for Youth | 3 month follow-up, 6 month follow-up and 2-year follow-up
  Self-report. Raw score range is 0-32 and higher scores indicate a worse outcome.
Difficulties in Emotion Regulation Skills | 3 month follow-up, 6 month follow-up and 2-year follow-up
  Self-report. Raw score range is 16-80 and higher scores indicate a worse outcome.
Compassionate Engagement and Action Scales - youth | 3 month follow-up, 6 month follow-up and 2-year follow-up
  Self-report. Raw score range is 0-270 and higher scores indicate a better outcome.
Strengths and Difficulties Questionnaire | 3 month follow-up, 6 month follow-up and 2-year follow-up
  Self-report. Raw score range is 0-40 and higher scores indicate a worse outcome.
EuroQualityOfLife - 5 Dimensions - Youth | 3 month follow-up, 6 month follow-up and 2-year follow-up
  Self-report. Raw score range is 5-15 and higher scores indicate a worse outcome.
Deliberate Self Harm Inventory | 3 month follow-up, 6 month follow-up and 2-year follow-up
  Self-report. Raw score range is 0-54 and higher scores indicate a worse outcome.
Montgomery Åsberg Depression Rating Scale - Youth | 3 month follow-up, 6 month follow-up and 2-year follow-up
  Self-report. Raw score range is 0-54 and higher scores indicate a worse outcome.
Suicidal Ideation Questionnaire | 3 month follow-up, 6 month follow-up and 2-year follow-up
  Self-report. Raw score range is 0-90 and higher scores indicate a worse outcome.
Emotional Breakthrough Inventory | 3 month follow-up, 6 month follow-up and 2-year follow-up
  Self-report. Raw score range is 0-100 and higher scores indicate a better outcome.
Patient-Reported Outcomes Measurement System (PROMIS), anger subscale | 3 month follow-up, 6 month follow-up and 2-year follow-up
  Self-report. Raw score range is 0-36 and higher scores indicate a worse outcome.
Patient-Reported Outcomes Measurement System (PROMIS), physical activity subscale | 3 month follow-up, 6 month follow-up and 2-year follow-up
  Self-report. Raw score range is 0-40 and higher scores indicate a better outcome.
Multiscale Dissociative Inventory | 3 month follow-up, 6 month follow-up and 2-year follow-up
  Self-report. Raw score range is 30-150 and higher scores indicate a worse outcome.
Negative experiences questionnaire | 3 month follow-up, 6 month follow-up and 2-year follow-up
  Self-report.
Paediatric side effect checklist | 3 month follow-up, 6 month follow-up and 2-year follow-up
  Self-report.
Heart rate variability | 3 month follow-up
  Bipolar Electrocardiography with no intervention after 15 min rest
Sleep registration | 6 week follow-up and 3 month follow-up.
  3-axial accelerometry-derived sleep efficiency/fragmentation/latency
Cortisol in hair | 3 month follow-up
  Average cortisol concentration in hair
Neuro-inflammation assay | 3 month follow-up
  Mesoscale micro-array on blood plasma
Growth factor assay | 3 month follow-up
  Mesoscale micro-array on blood plasma
Telomere length | 3 month follow-up
  Telomere length measured in peripheral blood mononuclear cells
Blood lipids | 3 month follow-up
  Standard lipid measures in blood plasma
Endocrine markers | 3 month follow-up
  Standard endocrine measures in blood serum
Avoidance and Fusion Questionnaire for Youth, mediation measure. | 6 week follow-up
  Self-rating. Mediation measure (TARA-arm participants only). Avoidance and Fusion Questionnaire for Youth. Raw score range is 0-32 and higher scores indicate a worse outcome.
Insomnia Severity Index, mediation measure. | 6 week follow-up
  Self-rating. Mediation measure (TARA-arm participants only). Insomnia Severity Index. Raw score range is 0-28 and higher scores indicate a worse outcome.
Difficulties in Emotion Regulation Skills, mediation measure | 6 week follow-up
  Self-rating. Mediation measure (TARA-arm participants only). Difficulties in Emotion Regulation Skills. Raw score range is 16-80 and higher scores indicate a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Henje, MD, PhD, Principal Investigator — Umeå Universitet
Locations (3):
- Sweden (3):
  - Ungdomshälsan/primary care, Umeå and Skellefteå, Västerbotten County
  - Barn och Ungdomspsykiatriska kliniken, Umeå, Skellefteå, and Lycksele, Västerbotten County
  - Barn och Ungdomspsykiatriska kliniken, Örnsköldsvik and Sundsvall, Västernorrland County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ekback E, Radmark L, Granasen G, Svarling R, Sorlin M, Schonbeck C, Henje E. Clinical effectiveness of training for awareness, resilience, and action for adolescents and young adults with depression: The pilot phase of a multicenter randomized controlled trial. Front Psychiatry. 2023 Mar 31;14:1130035. doi: 10.3389/fpsyt.2023.1130035. eCollection 2023. PMID 37065894
- [Derived] Ekback E, Granasen G, Svarling R, Blomqvist I, Henje E. Clinical Effectiveness of Training for Awareness Resilience and Action Online Compared to Standard Treatment for Adolescents and Young Adults With Depression: Study Protocol and Analysis Plan for a Pragmatic, Multi-Center Randomized Controlled Superiority Trial. Front Psychiatry. 2021 Oct 11;12:674583. doi: 10.3389/fpsyt.2021.674583. eCollection 2021. PMID 34707516

DOCUMENTS (1):
  • Study Protocol (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT04747340/Prot_001.pdf